CLINICAL TRIAL: NCT02791243
Title: A Within-subject, Randomized, Evaluator-blinded, Vehicle-controlled Study to Assess the Photosensitization Potential of Finasteride Cutaneous Solution(P-3074) in Human Subjects
Brief Title: Photosensitization Study in Androgenetic Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polichem S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PM1542
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Finasteride 0.25% (Experimental): approximately 0.2 ml of P-3074 (0.25% finasteride)
  Interventions: Drug: Finasteride 0.25%
- Placebo for Finasteride 0.25% (Placebo Comparator): approximately 0.2 ml of the vehicle cutaneous solution
  Interventions: Drug: Placebo for Finasteride 0.25%
- Negative Control (Other): approximately 0.2 ml of 0.9% aqueous NaCl
  Interventions: Drug: Negative Control

INTERVENTIONS:
Drug: Finasteride 0.25% — Cutaneous solution of finasteride 0.25%
  Other Names: P-3074
  Arms: Finasteride 0.25%
Drug: Placebo for Finasteride 0.25% — vehicle cutaneous solution of P-3074
  Other Names: vehicle cutaneous solution
  Arms: Placebo for Finasteride 0.25%
Drug: Negative Control — 0.9% aqueous NaCl
  Other Names: 0.9% aqueous NaCl
  Arms: Negative Control

SUMMARY:
This study evaluates the potential for induction of photosensitization by P-3074 0.25% finasteride cutaneous solution compared to that of placebo vehicle cutaneous solution and a negative control (0.9% sodium chloride, NaCl)

DETAILED DESCRIPTION:
Healthy male volunteers, drawn from the general population, will be treated with P-3074 solution, placebo vehicle control and 0.9% sodium chloride USP (negative control) by using 6 induction applications on the back area and Ultraviolet A (UVA)/Ultraviolet B (UVB) irradiations during the 3 week induction period, a 10 day rest period, and a challenge phase of a 24-hour patch application, UVA and UVB irradiation followed by evaluation of photosensitization over the subsequent 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 to 65.
2. Good general health, as assessed by verbal medical history and brief physical examination of the skin.
3. Fitzpatrick Skin Type I-IV, determined by interview at screening.
4. Willing to use a double-barrier methods (for example, a condom or a diaphragm plus spermicide) during sexual intercourse with a female partner while participating in the study.
5. Male subjects will need to confirm method and length of time for method of birth control for female partners.
6. Fully informed of the risks of entering the study and willing to provide written consent to enter the study.
7. Willing to follow study rules, which include: no sun exposure (for example, no swimming, sunbathing, or tanning beds), avoidance of activities that would cause excessive sweating, no use of lotions, creams, or oils on the back area
8. Must be willing not to change current brand of personal care products such as soaps, body washes, laundry detergent, body sprays, body spritzes, etc. while participating on the study.

Exclusion Criteria:

1. MED ≤ 2.5 SED for Fitzpatrick Skin Types I and II or MED ≤ 4.0 SED for Fitzpatrick Skin Types III and IV
2. Type I Insulin-dependent diabetes
3. Mastectomy for cancer involving removal of lymph nodes draining the test site.
4. Clinically significant skin diseases which may contraindicate participation, including psoriasis, eczema, atopic dermatitis, and active skin cancer.
5. Use of any photosensitizing medications or supplements, such as but not limited to sulfa drugs, tetracyclines, phenothiazines, thiazides, antiemetics and St. John's Wort.
6. Any medical conditions caused or affected by sunlight (UV), such as but not limited to solar urticarial and polymorphous light eruptions.
7. Active immunologic disorders.
8. Routine use of anti-inflammatory, immunosuppressive or antihistamine medications (81 mg aspirin is acceptable).
9. Participation in a patch test or soap chamber test within the past 4 weeks.
10. History of significant sensitivity or allergy to adhesive bandages, tapes, etc.
11. Use of finasteride (oral and/or topical), within 6 months prior to the screening visit.
12. Contraindications to finasteride therapy or intolerance of finasteride.
13. History of sensitivity to skin solution products.
14. Hair, tattoos, pigmentation, scars, moles or other conditions at the areas to be patched that may interfere with patch application, tolerability, or postapplication evaluations.
15. Participation in a clinical trial or receipt of an investigational medication within 4 weeks of the study.
16. Current treatment with allergy injections.
17. History of severe asthma.
18. Chronic or active liver disease [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5x upper limit of normal (ULN)]
19. Neutrophils < 1500 cells/mm3
20. Clinically significant chronic illness, which could place the subject at increased risk during participation or result in inappropriate dermal response during the study in the opinion of the Investigator.
21. History of alcohol or drug abuse within 1 year of the study.
22. Any condition the Investigator believes would interfere with the evaluation of the subject, or may put the subject at undue risk.
23. Judged by the investigator to be unsuitable for any reason.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06-27 (Actual)

PRIMARY OUTCOMES:
Potential for induction of photosensitization | from day 4 to day 42

CONTACTS AND LOCATIONS:
Overall Officials: Michael Carr, MD, Principal Investigator — Princeton Consumer Research Inc.
Locations (1):
- Princeton Consumer Research Inc., Chelmsford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No